CLINICAL TRIAL: NCT07249645
Title: Description of Return to Sport in Amateur Athletes Who Underwent Several Functional Tests (K-STARTS, Vertical Jumps and Soleus Muscle Strength) After Initial ACL Reconstruction.
Acronym: K-STARTS +
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01104-45
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
Keywords: Return To Sport ACL injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- K-STARTS + (Experimental): K-STARTS + arm involves following tests : K-STARTS, CMJ, DJ and soleus muscle strength measurement
  Interventions: Other: Physical tests

INTERVENTIONS:
Other: Physical tests — K-STARTS, CMJ, DJ, and soleus muscle strength measurement

SUMMARY:
ACL injuries are incapacitating for both professional and amateur athletes, with long-term repercussions on performance and return to sport (RTS).

Surgical reconstruction of the ACL is the main treatment option. Despite this, recurrence rates are high. Half of all recurrences occur within 8 months of reconstruction, and 70% within the first 6 months after RTS. Decision to RTS is therefore an important one, as returning too early can increase the risk of recurrence, while returning too late delays a return to pre-injury performance levels. As described by the Bern Consensus, RTS consists of three phases :

* Phase 1: Return to participation (RTp)
* Phase 2: Return to sport (RTS)
* Phase 3: Return to performance (RTP)

RTS decision must be based on multiple factors, including psychological, athletic and functional components, as well as specific nature of the patient's activities. However, few individual tests have been associated with a specific level of RTS. Furthermore, the majority of studies rely on subjective and non-objective assessments to determine whether the athlete has returned to their pre-injury level.

It would therefore be relevant to study the RTS time of patients who have performed a combination of several objective functional tests whose results could be complementary, in particular the K-STARTS, the CMJ, the DJ and the measurement of soleus muscle strength.

DETAILED DESCRIPTION:
ACL injuries are incapacitating for both professional and amateur athletes, with long-term repercussions on performance and return to sport (RTS). Only 60% of amateurs return to their pre-injury level of performance.

Surgical reconstruction of the ACL is the main treatment option. Despite this, recurrence rates are high (ranging from 17% to 40% depending on the population). Half of all recurrences occur within 8 months of reconstruction, and 70% within the first 6 months after RTS. The decision to RTS is therefore an important one, as returning too early can increase the risk of recurrence, while returning too late delays a return to pre-injury performance levels. As described by the Bern Consensus, RTS consists of three phases (Ardern et al. 2016):

* Phase 1: Return to participation (RTp)
* Phase 2: Return to sport (RTS)
* Phase 3: Return to performance (RTP)

RTS decision must be based on multiple factors, including psychological, athletic and functional components, as well as specific nature of the patient's activities. However, few individual tests have been associated with a specific level of RTS. Furthermore, the majority of studies rely on subjective and non-objective assessments to determine whether the athlete has returned to their pre-injury level. It would therefore be relevant to study the RTS time of patients who have performed a combination of several objective functional tests whose results could be complementary, in particular the K-STARTS, the CMJ, the DJ and the measurement of soleus muscle strength :

* The Knee Santy Athletic Return to Sport (K-STARTS) test, which includes psychological and functional assessments of the knee. The K-STARTS test consists mainly of horizontal jumps that assess the functional capabilities of the knee.
* A. Kotsifaki, et al. (2021) assessed the contribution of the knee joint during various horizontal and vertical jumping tasks. In particular, they reported a greater contribution of the knee during propulsion in vertical vs. horizontal jumps (34.1% vs. 12.9%, respectively) and, conversely, a greater contribution of the knee during landing in horizontal vs. vertical jumps (64.7% vs. 34.3%, respectively). Thus, the combination of vertical and horizontal jumps would allow for a functional assessment of the knee during the different phases of jumping. Counter-Movement Jump (CMJ) and drop jump (DJ) are the main types of vertical jumps recommended for functional assessment of the knee.
* Measurement of soleus muscle strength. Recent studies have shown a decrease in the contribution of the soleus muscle during propulsion and landing in horizontal and vertical jumps in subjects with ACL injury.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged between ≥ 18 and ≤ 30 years old
* Amateur athlete with a Tegner score ≥ 5
* Patient with primary ACL reconstruction dating back 6 months
* Patients with ACL damage in one knee only
* Patients who have undergone an isokinetic strength test with results that do not contraindicate functional testing
* Patients affiliated with or covered by a social security scheme
* French-speaking patients who have signed an informed consent form

Exclusion Criteria:

* Patients treated for bilateral ACL reconstruction
* Patients who are professional athletes or compete at a national level
* Patients with severe associated disorders (neurological, connective tissue, congenital diseases)
* Patients with multiple ligament defects or associated osteotomy
* Patients already included in another study
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Return to sport | 18 months
  This is time period (in months) between surgery and:
  * The date of return to sport (phase 2) for patients who resumed sport
  * The end of follow-up (timepoint date/date of death/date of loss of contact) for patients who did not resume sport

IPD SHARING:
Plan to Share IPD: No